CLINICAL TRIAL: NCT07227987
Title: Cognitive Rehabilitation for Treatment of Anger in Veterans With TBI (Traumatic Brain Injury) and PTSD (Post-traumatic Stress Disorder)
Brief Title: Cognitive Rehabilitation for Treatment of Anger in Veterans With TBI and PTSD
Acronym: CALM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00118644; CDMRP-TP240244 (Other: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2025-11-11; First posted 2025-11-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury (TBI); Posttraumatic Stress Disorder (PTSD)
Keywords: Traumatic Brain Injury (TBI); Posttraumatic stress Disorder (PTSD); Mobile app; Veterans
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participant dyads will be randomized to either Cognitive Rehabilitation (n=50) or Psychoeducation (n=50).
Who Masked: Outcomes Assessor
Masking Description: To maintain blinding of the 3-month and 6-month interviewers to participants' treatment assignments: 1) The first interviewer will collect study equipment at follow-ups; 2) A different interviewer will handle the 3- and 6-month interviews; 3) Participants will be instructed not to discuss their intervention details during follow-up; and 4) The participant tracking database will be protected, accessible only to study coordinators who conducted the baseline assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CALM (Cognitive Apps for Life Management) (Experimental)
  Interventions: Other: CALM (Cognitive Apps for Life Management)
- Psychoeducation (Active Comparator)
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Other: CALM (Cognitive Apps for Life Management) — GMT + content-free cueing + n-back task
  1. Goal Management Training: cognitive strategies to help Veterans improve goal-setting, planning, and self-monitoring in real world contexts.
  2. Content-free cueing: intermittent prompts to conduct an "executive review" received four times daily on participant's smartphone, aimed to help improve goal-directed actions and self-monitoring of one's behavior.
  3. N-back task: Veterans practice an n-back task via the mobile app, which aims to improve working memory and inhibitory control.
  Arms: CALM (Cognitive Apps for Life Management)
Other: Psychoeducation — Brain Health Training + Concussion Coach app Participants in the active control group will receive psychoeducational material as part of the "Brain Health Training" used as a control in cognitive rehabilitation and Goal Management Training (GMT). Veterans will also use "Concussion Coach," a VA and DoD app providing resources on TBI and cognitive functioning tips.
  Arms: Psychoeducation

SUMMARY:
This randomized clinical trial will enroll 100 Veteran-family/friend dyads to test the efficacy of CALM in treating anger in TBI and PTSD. The investigators hypothesize that compared to an active control group, Veterans randomized to the CALM group will demonstrate:

* Significantly larger decreases in anger dysregulation, impulsivity, and executive dysfunction.
* Significantly larger improvements in social and adaptive functioning including less aggression.
* Significantly larger reduction in PTSD symptoms and suicidal ideation.

The study targets Veterans who experience difficulties with anger and impulsivity due to TBI and PTSD. These issues are common, with up to 38% of Veterans with TBI also having PTSD. These conditions often make it challenging for Veterans to control their emotions and interact successfully in social and work settings. Our research will test the CALM (Cognitive Applications for Life Management) mobile app, which helps Veterans manage their goals, remember important tasks, and improve their attention. Initial tests of CALM have shown it can reduce levels of anger and related issues in Veterans. The investigators will conduct a study with 100 pairings of Veterans and a family member or friend. These pairs will be randomly assigned to one of two groups: one using the CALM mobile platform and the other receiving brain health education. Both groups will use their assigned intervention for three months and will receive support through videoconference calls at the beginning, middle, and end of the program.

DETAILED DESCRIPTION:
In military populations, traumatic brain injury (TBI) and posttraumatic stress disorder (PTSD) frequently co-occur, with prevalence rates indicating that 34% to 38% of Service members and Veterans diagnosed with TBI also meet criteria for PTSD. Brain areas affected by TBI are implicated in PTSD, particularly in the frontal lobe involved in executive function and emotional and behavioral regulation. Veterans with TBI and PTSD often face challenges such as biological dysregulation secondary to brain injury, including difficulty managing anger, diminished inhibitory control, and increased aggression and suicide.

Interventions aimed at effectively addressing these adverse outcomes are limited, however. As noted in the Centers for Disease Control (CDC) report cited in the current CDMRP Program Announcement, PTSD-focused and mind-body treatments for anger have proven ineffective. For that reason, there is a critical imperative to discover other methods to reduce anger and impulsivity in Service members and Veterans with TBI and PTSD. Given neural mechanisms implicated in TBI and PTSD, an alternative approach to directly treat anger is to improve executive function itself. The Supervisory Attentional System (SAS) conceptualizes executive function as involving inhibition, attention, self-monitoring, and planning. These processes, along with emotional regulation, are key targets of a theory-based cognitive rehabilitation of executive function.

To improve executive function in TBI, research supports use of multiple approaches to optimize self-monitoring, emotion regulation, and self-control. One evidence-based intervention for executive function in TBI is goal management training (GMT). GMT trains individuals with TBI to set self-directed personal goals (e.g., work, school, fitness), break complex tasks into steps, and monitor attention to gain cognitive control. Multiple systematic reviews show GMT improves outcomes such as emotional regulation and social functioning, including among Veterans and non-Veterans with co-occurring TBI and PTSD. Another related approach involves external cues which can be used to encourage individuals with TBI to practice goal-directed behavior in real-world situations by prompting an "executive review" (e.g., asking oneself "What is the goal of what I'm doing right now? What are the steps to that goal? Am I paying attention to each step?"). Research shows cueing and conducting executive reviews is associated with fewer functional limitations in individuals with TBI. This content-free cueing involving several daily reminders helps apply goal-oriented behaviors in daily life, leading to better emotional regulation and social functioning after brain injury.

Finally, attention training has also been shown to be effective in reducing function limitations in TBI. The n-back task in particular has been used to increase attentional control, inhibition, and working memory by training conscious and deliberate use of strategies to effectively allocate attentional resources and manage the rate of information received during task completion, with recent studies showing working memory interventions in general, and n-back training specifically, change neural pathways and improve attentional control. All three (GMT, content free-cuing, and the n-back task) can be implemented via mobile health technology, extending cognitive rehabilitation from the clinic to the home. Optimal rehabilitation also capitalizes on an individual's social support network, particularly relevant for successful reintegration after military service for Veterans with TBI and PTSD. The investigators have found links between Veterans' social support and improved treatment engagement, reduced violence, and reduced suicide risk.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Veterans

* U.S. Veteran who served in one of the military branches (Army, Navy, Marines, Air Force, or Coast Guard) since 9/11/01
* Meets criteria for TBI
* Meets criteria for PTSD or subthreshold PTSD
* Reports anger problems began after their head injury
* Reports current problems with cognitive function
* At least 18 years old
* Fluent and literate in English
* Able to provide voluntary, informed consent to participate.

Inclusion Criteria for Family members or Friends:

* Over age 18;
* Family member/friend of Veteran who served in one of the military branches (Army, Navy, Marines, Air Force, National Guard) post-9/11 and who meets TBI and PTSD inclusion criteria
* Fluent and literate in English
* Able to provide voluntary, informed consent to participate.

Exclusion Criteria:

* Does not own a smartphone.
* Does not have a trusted support person, e.g., spouse, family member, or friend for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dimensions of Anger (DAR7) | Baseline, 3 months, 6 months
  The Dimensions of Anger Reactions-7 (DAR-7) measures an individual's propensity to experience, express, and manage anger. It consists of 7 items assessing anger frequency, intensity, duration, and the impact on behavior and relationships.
Barratt Impulsiveness Scale-11 (BIS-11) | Baseline, 3 months, 6 months
  Barratt Impulsiveness Scale-11 is designed to measure impulsivity as a personality trait. It includes 30 items that assess three key dimensions: attentional impulsiveness (lack of focus), motor impulsiveness (acting without thinking), and non-planning impulsiveness (lack of forethought).
Delis-Kaplan Executive Function System (D-KEFS) | Baseline, 3 months, 6 months
  The Delis-Kaplan Executive Function System (D-KEFS) is a comprehensive battery of neuropsychological tests designed to assess a wide range of executive functions, such as problem-solving, cognitive flexibility, inhibition, and planning. It includes nine stand-alone subtests that evaluate higher-order thinking skills involved in goal-directed behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Elbogen, Principal Investigator — Duke University
Locations (1):
- Duke University School of Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The Federal Interagency Traumatic Brain Injury Research (FITBIR) informatics system was developed to share data across the entire TBI research field and to facilitate collaboration between laboratories, as well as interconnectivity with other informatics platforms.
Time Frame: Data uploaded to FITBIR on a quarterly basis, per Data Sharing Policy.
Access Criteria: All links with participants identity will be removed from the data before they are shared. Only de-identified data which do not include anything that might directly identify participants will be shared with FITBIR users and the general scientific community for research purposes.